CLINICAL TRIAL: NCT00058539
Title: A Phase II, Open-Label, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Omnitarg (Pertuzumab) in Subjects With Castration-Resistant Prostate Cancer
Brief Title: Safety and Efficacy Study of Pertuzumab to Treat Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOC2682g; NCT00066755 (obsolete NCT alias)
Record Dates: First submitted 2003-04-08; First posted 2003-04-09 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pertuzumab

INTERVENTIONS:
Drug: rhuMAb 2C4 (pertuzumab)

SUMMARY:
The purpose of this study is to evaluate safety and efficacy of Omnitarg (Pertuzumab) on cancerous lesions in men with castration-resistant (hormone-refractory) prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age >= 18 years old
* Histologically documented adenocarcinoma of the prostate, clinically refractory or resistant to hormone therapy, as assessed by progression following at least one hormonal therapy (orchiectomy or luteinizing hormone-releasing hormone [LHRH] agonist). Subjects must have documented progression following hormonal therapy withdrawal of >= 4 weeks duration; nilutamide and bicalutamide require 6 weeks withdrawal.
* Progression of disease after one prior chemotherapy regimen (which must have been taxane-based) for CRPC. Progression is defined as at least one of the following: A minimum of three consecutive serum PSA measurements obtained >= 14 days apart and all within 3 months, with progressively increasing values for two consecutive measurements. The latest value must be obtained within the screening period and must be >= 5 ng/mL; or progression of measurable disease, as defined by RECIST; or progression of bone disease, as defined by the appearance of one or more new bone lesions
* Orchiectomy, or castrate levels of testosterone maintained by LHRH agonist <70 ng/mL
* Life expectancy >= 12 weeks
* ECOG performance status of 0 or 1
* Granulocyte count of >= 1500/mL, platelet count of >= 75,000/mL and hemoglobin of >= 9 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbopoeitin [Aranesp] is permitted)
* Serum bilirubin less than or equal to the upper limit of normal (ULN), unless due to Gilbert's disease, and alkaline phosphatase, AST, and ALT <= 2.5 x ULN (ALT, AST, and alkaline phosphatase <= 5 x ULN for subjects with liver metastases; no alkaline phosphatase upper limit for subjects with bone metastases)
* Serum creatinine <= 1.5 x ULN
* International normalized ratio (INR) <1.5 and activated partial thromboplastin time (aPTT) <1.5 x ULN (except for subjects receiving warfarin)
* Willing to complete serial PROSQOLI/PPI evaluations and serial diaries of analgesic use (if necessary)

Exclusion Criteria:

* Prior chemotherapy, radiotherapy, therapeutic radionucleotide or immunotherapy within 4 weeks of Day 1 (the day of the first rhuMAb 2C4 dose). Flutamide therapy, or other second line hormonal therapies should be withdrawn >= 4 weeks prior to Day 1. Bicalutamide and nilutamide therapy should be withdrawn >= 6 weeks prior to starting study medication.
* Prior treatment with HER2 pathway inhibitors (e.g., Herceptin [Trastuzumab], Iressa [gefitinib], Tarceva [erlotinib hydrochloride], C225, CI1033, and TAK165)
* Treatment with other experimental anticancer agents within 4 weeks prior to Day 1
* Prior history or clinical evidence of central nervous system or brain metastases
* Ejection fraction, determined by ECHO, <50%
* Uncontrolled hypercalcemia (>11.5 mg/dL)
* Prior exposure of >360 mg/m2 doxorubicin, >120 mg/m2 mitoxantrone, or >90 mg/m2 idarubicin
* Ongoing corticosteroid treatment, except for subjects who are on stable doses of <20 mg of prednisone daily (or equivalent), or who are taking corticosteroids for reasons unrelated to prostate cancer
* History of other malignancies within 5 years prior to Day 1, except for adequately treated basal or squamous cell skin cancer
* History of serious systemic disease, including active infection, uncontrolled hypertension (diastolic blood pressure >100 mmHg on two consecutive occasions), unstable angina, congestive heart failure, or myocardial infarction within 6 months prior to Day 1, or unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation, paroxysmal supraventricular tachycardia, or controlled hypertension are eligible)
* Ongoing liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus infection
* Major surgery or significant traumatic injury within 3 weeks prior to Day 1
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk for treatment complications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-04; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab: All the participants received a loading dose of 840 milligrams (mg) of pertuzumab on Day 1 of Cycle 1, followed by 420 mg on Day 1 of each subsequent 21-day cycle. Pertuzumab was administered as an intravenous (IV) infusion every 3 weeks for up to 1 year (17 cycles) for participants who showed no evidence of progression. Participants with evidence of disease progression could have continued pertuzumab therapy, at the discretion of the investigator, if they had improvement in pain without an increase in narcotic use and if they had no other therapeutic options.
Period: Overall Study
Arm/Group | Pertuzumab
Started | 42
Completed | 0
Not Completed | 42
Not completed — Disease progression | 24
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 9
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All the participants who received at least 1 dose of study drug were included in the analysis.
Groups:
- Pertuzumab: All the participants received a loading dose of 840 mg of pertuzumab on Day 1 of Cycle 1, followed by 420 mg on Day 1 of each subsequent 21-day cycle. Pertuzumab was administered as an IV infusion every 3 weeks for up to 1 year (17 cycles) for participants who showed no evidence of progression. Participants with evidence of disease progression could have continued pertuzumab therapy, at the discretion of the investigator, if they had improvement in pain without an increase in narcotic use and if they had no other therapeutic options.
Arm/Group | Pertuzumab
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Confirmed Response of Complete Response (CR) or Partial Response (PR) Based on Response Evaluation Criteria in Solid Tumors (RECIST) and Prostate Specific Antigen (PSA) Response Rate Based on Bubley Criteria
Description: Response by tumor measurement occurred if there was documented and confirmed CR or PR. Response was assessed by both the RECIST and by PSA levels measurement, based on measurable or non-measurable disease at baseline. Per RECIST, CR: disappearance of all target and non-target lesions and normalization of tumor marker level; PR: at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. A PSA response was defined as a PSA decline of greater than or equal to (≥) 50%, which had to be confirmed by a second PSA value at least 4 weeks later.
Time Frame: Screening, Day 1 of Cycles 1-17, and at 30 days after the last dose of pertuzumab
Population: Efficacy analysis population: All participants who received at least 1 dose of study drug and either underwent at least 1 postbaseline assessment of response or died within 30 days after the last study treatment before any evaluation of response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 30
percentage of participants | 0.0 [0.0 to 0.0]

2. Primary Outcome: Kaplan Meier Estimate of Percentage of Participants With Disease Progression at 3 Months
Description: Per RECIST, disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of 1 or more new lesions, and/or unequivocal progression of existing non-target lesions.
Time Frame: 3 months
Population: Efficacy analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 30
percentage of participants | 80

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death (Progression Free Survival [PFS])
Description: PFS was defined as the time from the first day of study drug treatment to the time of documented disease progression or death, whichever came first. Participants who were lost to follow-up or who had not progressed at the time of study completion or early termination were censored at the date of last tumor assessment. The percentage of participants experiencing disease progression or death was calculated as the number of participants with an event divided by the number of participants analyzed, multiplied by 100.
Time Frame: Screening, Day 1 of Cycles 1-17, and at 30 days after the last dose of pertuzumab
Population: Efficacy analysis population. Five participants were censored for this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 30
percentage of participants | 83.3

4. Secondary Outcome: Median Time of PFS
Description: PFS was defined as the time from the first day of study drug treatment to the time of documented disease progression or death, whichever came first. Participants who were lost to follow-up or who had not progressed at the time of study completion or early termination were censored at the date of last tumor assessment.
Time Frame: Screening, Day 1 of Cycles 1-17, and at 30 days after the last dose of pertuzumab
Population: Efficacy analysis population. Five participants were censored for this analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pertuzumab
Number analyzed (Participants) | 30
weeks | 9.6 [9.1 to 11.1]

5. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the initial CR or PR to the time of disease progression.
Time Frame: Screening, Day 1 of Cycles 1-17, and at 30 days after the last dose of pertuzumab
Population: No participants experienced either CR or PR.
Arm/Group | Pertuzumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Participants Who Progressed at 3, 6 and 9 Months
Description: Per RECIST, disease progression was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started or the appearance of 1 or more new lesions, and/or unequivocal progression of existing non-target lesions. Percentage of participants who were free from disease progression was calculated by subtracting the number of participants with disease progression at that time point from the total population at risk of disease progression, multiplied by 100.
Time Frame: 3, 6, and 9 months
Population: Efficacy analysis population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab
Number analyzed (Participants) | 30
percentage of participants
  % of participants progressed at 3 months | 66.7
  % of participants progressed at 6 months | 80.0
  % of participants progressed at 9 months | 83.3

7. Secondary Outcome: Serum Concentrations of Pertuzumab
Time Frame: Assessed at pre-dose, 15-minutes postdose on Day 1 (Cycle 1), Day 22 (Cycle 2), Day 43 (Cycle 3), Day 85 (Cycle 5), and Day 169 (Cycle 9); pre-dose on Day 253 (Cycle 13), and on Days 8, 15, 29 and 36
Population: Pharmacokinetic evaluable participants
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Pertuzumab
Number analyzed (Participants) | 40
micrograms per milliliter (µg/mL)
  Day 1, 15 minutes postdose (n=38) | 254.71 (46.85)
  Day 8 (n=39) | 97.51 (25.93)
  Day 15 (n=38) | 69.23 (19.13)
  Day 22 pre-dose (n=33) | 52.41 (15.23)
  Day 22, 15 minutes postdose (n=31) | 175.87 (34.70)
  Day 29 (n=30) | 88.17 (27.83)
  Day 36 (n=32) | 67.45 (21.46)
  Day 43 pre-dose (n=26) | 53.09 (19.45)
  Day 43, 15 minutes postdose (n=23) | 176.17 (32.43)
  Day 85 pre-dose (n=5) | 67.36 (23.66)
  Day 85, 15 minutes postdose (n=4) | 199.50 (35.07)
  Day 169 pre-dose (n=3) | 75.97 (49.41)
  Day 169, 15 minutes postdose (n=3) | 207.67 (71.70)
  Day 253 pre-dose (n=1) | 40.7 (NA) — Standard deviation was not analyzed for single participant.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline until up to 30 days after the last dose of pertuzumab.
Arm/Group | Pertuzumab
Serious Adverse Events (participants affected / at risk) | 11/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab (N=41)
Constipation (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Ureteric obstruction (Renal and urinary disorders) | 2
Bilateral hydronephrosis (Renal and urinary disorders) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Tachycardia (Cardiac disorders) | 1
Pain (General disorders) | 1
Stent occlusion (Injury, poisoning and procedural complications) | 1
Troponin t increased (Investigations) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuropathy (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab (N=41)
Diarrhoea (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 14
Oedema peripheral (General disorders) | 8
Mucosal inflammation (General disorders) | 6
Pain (General disorders) | 6
Asthenia (General disorders) | 5
Pyrexia (General disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Ejection fraction decreased (Investigations) | 12
Activated partial thromboplastin time prolonged (Investigations) | 3
Prothrombin time prolonged (Investigations) | 3
Weight decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 11
Decreased appetite (Metabolism and nutrition disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 3
Hypoaesthesia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Dysuria (Renal and urinary disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.